The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for a single centre, open label, one sequence, cross-over study to evaluate the effect of itraconazole on the pharmacokinetics of single inhaled doses of nemiralisib in healthy volunteers.

Compound Number : GSK2269557

Effective Date : 12-APR-2018

## Description:

 The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206874.

- This RAP is intended to describe the final analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

## RAP Author(s):

| Approver | Date | Approval Method |
|---|---|---|
| PPD | 20 MAD 2019 | NI/A |
| Statistics Leader (Respiratory Clinical Statistics) | 20-MAR-2018 | N/A |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Manager (Respiratory Clinical Pharmacology<br>Modelling and Simulation) | 21-MAR-2018 | Electronically<br>within C.A.R.S.<br>system |
| Clinical Program Lead (Clinical Pharmacology<br>Science and Study Operations) | 21-MAR-2018 | Electronically<br>within C.A.R.S.<br>system |
| Physician (Respiratory) | 12-APR-2018 | Email |
| Programming Manager (Respiratory Clinical Programming) | 20-MAR-2018 | Electronically<br>within C.A.R.S.<br>system |
| Data Quality Lead (Respiratory Data<br>Management) | 26-MAR-2018 | Electronically<br>within C.A.R.S.<br>system |
| Medical Director (Global Clinical Safety & Pharmacovigilance) | 10-APR-2018 | Electronically<br>within C.A.R.S.<br>system |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Director (Respiratory Clinical Statistics) | 20-MAR-2018 | Electronically<br>within C.A.R.S.<br>system |
| Manager (Respiratory Clinical Programming) | 23-MAR-2018 | Electronically<br>within C.A.R.S.<br>system |

## **TABLE OF CONTENTS**

| | | P | AGE |
|---|---|---|---|
| 1. | INTRODU | ICTION | 5 |
| 2. | SUMMAR | Y OF KEY PROTOCOL INFORMATION | 5 |
| ۷. | | nanges to the Protocol Defined Statistical Analysis Plan | |
| | | udy Objective(s) and Endpoint(s) | |
| | | udy Objective(s) and Enapoint(s)udy Design | |
| | | atistical Hypotheses / Statistical Analyses | |
| 3. | | O ANALYSES | 8 |
| | | erim Analyses | |
| | 3.2. Fir | nal Analyses | 8 |
| 4. | | S POPULATIONS | |
| | 4.1. Pro | otocol Deviations | 9 |
| 5. | | ERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | TIONS | |
| | | udy Treatment & Sub-group Display Descriptors | |
| | | seline Definitions | |
| | | ultiple Comparisons and Multiplicityher Considerations for Data Analyses and Data Handling | 10 |
| | | onventions | 11 |
| 6. | CTLIDV D | OPULATION ANALYSES | 10 |
| Ο. | | verview of Planned Study Population Analyses | |
| | 0.1. | civion of rialimod clady repulation randings committee in the committee of | |
| 7. | PHARMA | COKINETIC ANALYSES | 13 |
| | 7.1. Pri | imary Pharmacokinetic Analyses | 13 |
| | 7.1 | 1.1. Endpoint / Variables | 13 |
| | | 7.1.1.1. Drug Concentration Measures | 13 |
| | | 7.1.1.2. Derived Pharmacokinetic Parameters | 13 |
| | 7.1 | 1.2. Summary Measure | 13 |
| | 7.1 | 1.3. Population of Interest | |
| | 7.1 | 1.4. Strategy for Intercurrent (Post-Randomization) Events | 13 |
| | 7.1 | 1.5. Statistical Analyses / Methods | |
| | | 7.1.5.1. Statistical Methodology Specification | 14 |
| | 7.2. Se | condary Pharmacokinetic Analyses | 15 |
| | 7.2 | 2.1. Endpoint / Variables | 15 |
| | | 7.2.1.1. Drug Concentration Measures | 15 |
| | | 7.2.1.2. Derived Pharmacokinetic Parameters | 15 |
| | 7.2 | 2.2. Summary Measure | 15 |
| | 7.2 | 2.3. Population of Interest | 15 |
| | 7.2 | 2.4. Statistical Analyses / Methods | 16 |
| 8. | SAFETY A | ANALYSES | 17 |
| | | Iverse Events Analyses | |
| | | Iverse Events of Special Interest Analyses | |
| | | inical Laboratory Analyses | |
| | | her Safety Analyses | |

| 9. | | PHARMACOKINETIC (POPPK)/ PHYSIOLOGICALLY-BASED PK (PBPK) | |
|---|---|---|---|
| | | 'SES | |
| | 9.1. | Statistical Analyses / Methods | 18 |
| 10. | REFER | RENCES | 19 |
| 11. | APPEN | NDICES | 20 |
| | 11.1. | Appendix 1: Schedule of Activities | |
| | | 11.1.1. Protocol Defined Schedule of Events | |
| | 11.2. | Appendix 2: Study Phases and Treatment Emergent Adverse | |
| | | Events | 25 |
| | | 11.2.1. Study Phases for Concomitant Medication | |
| | | 11.2.2. Treatment Emergent Flag for Adverse Events | |
| | 11.3. | Appendix 3: Data Display Standards & Handling Conventions | |
| | | 11.3.1. Reporting Process | |
| | | 11.3.2. Reporting Standards | 26 |
| | | 11.3.3. Reporting Standards for Pharmacokinetic | 27 |
| | 11.4. | Appendix 4: Derived and Transformed Data | 28 |
| | | 11.4.1. General | 28 |
| | | 11.4.2. Study Population | |
| | | 11.4.3. Safety | |
| | 11.5. | Appendix 5: Reporting Standards for Missing Data | |
| | | 11.5.1. Premature Withdrawals | |
| | | 11.5.2. Handling of Missing Data | |
| | | 11.5.2.1. Handling of Missing and Partial Dates | |
| | 11.6. | Appendix 6: Values of Potential Clinical Importance | 32 |
| | | 11.6.1. Laboratory Values | |
| | | 11.6.2. ECG | |
| | | 11.6.3. Vital Signs | |
| | 11.7. | Appendix 7: Abbreviations & Trade Marks | |
| | | 11.7.1. Abbreviations | |
| | 44.0 | 11.7.2. Trademarks | |
| | 11.8. | Appendix 8: List of Data Displays | |
| | | 11.8.1. Data Display Numbering | |
| | | 11.8.2. Mock Example Shell Referencing | |
| | | 11.8.3. Deliverables | |
| | | 11.8.4. Study Population Tables | |
| | | 11.8.5. Pharmacokinetic Tables | |
| | | 11.8.6. Pharmacokinetic Figures | |
| | | 11.8.7. Safety Tables | |
| | | 11.8.8. ICH Listings | |
| | 11 0 | 11.8.9. Non-ICH Listings | טו |
| | 1 1.J. | ADDUTUIA J. LAGITIDIE MUUR OTIETIS IUI DALA DISDIAVS | UU |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 206874:

| Revision Chronology | | |
|---------------------|-------------|----------|
| 2017N347248_00 | 12-DEC-2017 | Original |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 12/DEC/2017).

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To characterize the effect of repeat oral dosing of itraconazole on the pharmacokinetics of a single inhaled dose of GSK2269557 (nemiralisib) in healthy subjects. Secondary Objectives | <ul> <li>AUC(0-∞)</li> <li>AUC(0-t)</li> <li>Cmax</li> <li>Tmax</li> <li>t<sub>1/2</sub></li> <li>Secondary Endpoints</li> </ul> |
| To investigate the safety and tolerability of single inhaled dose of nemiralisib, when dosed alone and concomitantly with itraconazole, in healthy subjects. | <ul> <li>Adverse events (AE),</li> <li>Clinical laboratory values,</li> <li>Vital signs,</li> <li>Electrocardiogram (ECG) and</li> <li>Spirometry.</li> </ul> |
| To investigate the pharmacokinetics of itraconazole and hydroxy itraconazole when coadministered with nemiralisib. | <ul> <li>AUC(0-∞)</li> <li>AUC(0-t)</li> <li>Cmax</li> <li>tmax</li> <li>t<sub>1/2</sub></li> </ul> |

 $AUC(0-\infty)$  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time, AUC(0-t): Area under the plasma concentration versus time curve from time zero to t, Cmax: maximum observed plasma concentration, tmax: time to Cmax,  $t_{1/2}$ : Terminal phase half-life.

## 2.3. Study Design



## 2.4. Statistical Hypotheses / Statistical Analyses

This study is designed to characterise the effect of repeat oral dosing of itraconazole on the pharmacokinetics of a single inhaled dose of nemiralisib in healthy participants. In particular, a comparison will be made between:

• The exposure of nemiralisib administered alone and the exposure of nemiralisib co-administered following repeat doses of itraconazole.

For AUC( $0-\infty$ ) and Cmax, point estimates and corresponding two-sided 90% confidence intervals (CIs) will be constructed for the ratio of the geometric means. No formal hypotheses will be tested.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

Following the availability of PK data prior to DBF, a preliminary assessment of unblinded PK data will be performed by CPMS using nominal timepoints. This assessment will be for internal decision making only, will not be formally reported and SAC deliverables will supersede any such output.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants screened and for whom a record exists on the study database. | Screening Status/Screening Failures |
| Enrolled | <ul> <li>All participants who passed screening and entered the study. Included are: run-in failures; and participants who took treatment.</li> <li>Note screening failures and participants screened but never enrolled into the study are excluded from the Enrolled population as they did not enter the study.</li> </ul> | <ul><li>Summary of Study<br/>Populations</li><li>Summary of Age<br/>Ranges</li></ul> |
| Safety | <ul> <li>All participants enrolled in the study, who took at least one dose of study treatment.</li> <li>Participants will be analysed according to the treatment they actually received.</li> <li>Note: Participants who were not assigned treatment but received at least one dose of study treatment should be listed.</li> </ul> | <ul><li>Other Study<br/>Population</li><li>Safety</li></ul> |
| Pharmacokinetic (PK) | <ul> <li>All participants enrolled in the study who took at least 1 dose of nemiralisib and for whom a nemiralisib pharmacokinetic sample was obtained and analysed.</li> <li>Participants will be analysed according to the treatment they received.</li> </ul> | • PK |

Refer to Appendix 8: List of Data Displays which details the population used for each display.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised in the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions |
|---------------------------------------------|
| Data Displays for Reporting |
| Description Order in TLF |
| NEMI 100mcg SD Alone 1 |
| NEMI 100mcg SD with Itraconazole 200mg RD 2 |

Treatment comparisons will be displayed using the descriptors as follows:

• NEMI 100mcg SD with Itraconazole 200mg RD vs. NEMI 100mcg SD Alone

## 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions below) the baseline value will be the latest pre-dose assessment with a non-missing value, for the relevant period, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. Note that baseline for FEV1 is defined as the screening visit in the protocol; however it is not required in any data displays so is not included here.

| Parameter | Study Assessments Considered as Baseline | | Baseline Used in Data<br>Display |
|---|---|---|---|
| | Screening | Day 1 (Pre-Dose)<br>[Periods 1 and 2] | |
| Safety | | | |
| Vital Signs | X <sup>1</sup> | Х | Day 1 predose for the relevant period |
| ECG | X <sup>1</sup> | Х | Day 1 predose for the relevant period |

<sup>[1]</sup> Triplicate

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

## 5.3. Multiple Comparisons and Multiplicity

No adjustments for multiplicity will be made.

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the following appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| 11.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 11.4 | Appendix 4: Derived and Transformed Data |
| 11.5 | Appendix 5: Reporting Standards for Missing Data |
| 11.6 | Appendix 6: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 8: List of Data Displays.

#### 7. PHARMACOKINETIC ANALYSES

## 7.1. Primary Pharmacokinetic Analyses

#### 7.1.1. Endpoint / Variables

#### 7.1.1.1. Drug Concentration Measures

Nemiralisib drug concentration data will be displayed as detailed in Appendix 3: Data Display Standards & Handling Conventions (Section 11.3.3 Reporting Standards for Pharmacokinetic).

#### 7.1.1.2. Derived Pharmacokinetic Parameters

Nemiralisib pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. The nemiralisib pharmacokinetic parameters listed below will be determined from the plasma concentration-time data, as data permit.

| Parameter | Parameter Description |
|---|---|
| AUC(0-∞) | Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite |
| , | time. $AUC(0-\infty) = AUC(0-t) + C(t)/\lambda z$ . |
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable |
| | concentration |
| %AUCex | Percentage of AUC(0-∞) obtained by extrapolation |
| Cmax | Maximum observed plasma concentration |
| tmax | Time to Cmax |
| t <sub>½</sub> | Apparent terminal half-life. $t_{1/2} = \ln 2/\lambda z$ |

#### NOTES:

- Additional parameters may be included as required.
- λz is the terminal phase rate constant.

#### 7.1.2. Summary Measure

The parameters for treatment comparisons are AUC(0- $\infty$ ), AUC(0-t), Cmax, tmax and  $t_{\frac{1}{2}}$  for nemiralisib.

#### 7.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

Two intercurrent events have been identified and will be handled by differing strategies:

- A *while on treatment* strategy will be employed for treatment discontinuation from nemiralisib (i.e. treatment discontinuation prior to dosing with nemiralisib on day 5 of period 2).
- A *hypothetical* strategy will be employed for treatment discontinuation from itraconazole (i.e. treatment discontinuation after dosing with nemiralisib on day 5 of period 2).

## 7.1.5. Statistical Analyses / Methods

Details of the planned displays for nemiralisib PK data are provided in Appendix 8: List of Data Displays, and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. Subjects with greater than 20% extrapolated AUC(0-∞) will be flagged.

## 7.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses for nemiralisib will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles). If  $AUC(0-\infty)$  is not calculable for more than 50% of subjects in the PK population in each period, AUC (0-t) will also be analysed for nemiralisib as described below.

## **Endpoint / Variables**

- AUC(0-∞) for nemiralisib
- Cmax for nemiralisib

#### Model Specification

- The parameters AUC(0-∞) and Cmax will be log<sub>e</sub> transformed and analysed separately using mixed effects models.
- Treatment Group will be fitted as a fixed effect and subject as a random effect.
- The MIXED procedure in SAS will be used with the following options:-
  - The Kenward and Roger method for approximating the denominator degrees of freedom to correct for bias in the estimated variance-covariance.
- Nemiralisib co-administered with itraconazole will be compared to nemiralisib administered alone.

#### **Model Checking & Diagnostics**

Distributional assumptions underlying the models used for analysis will be examined by
obtaining box plots and normal probability plots of the studentised residuals and plots of the
residuals versus the fitted values (i.e. checking the normality assumption and constant
variance assumption of the model respectively) to gain confidence that the model assumptions
are reasonable.

#### **Model Results Presentation**

- For each PK parameter:-
  - Adjusted geometric means and 90% confidence intervals (CI) for each treatment group and standard error (log<sub>e</sub> scale).

- Point estimates and associated two-sided 90% confidence intervals for the ratio of nemiralisib co-administered with itraconazole to nemiralisib administered alone (obtained by back-transforming estimates and 90% CIs for the treatment differences from the statistical model on the loge scale) and standard error (loge scale).
- The mean squared error (MSE) will also be presented.

## 7.2. Secondary Pharmacokinetic Analyses

## 7.2.1. Endpoint / Variables

#### 7.2.1.1. Drug Concentration Measures

Itraconazole and hydroxy-itraconazole drug concentration data will be displayed as detailed in Appendix 3: Data Display Standards & Handling Conventions (Section 11.3.3 Reporting Standards for Pharmacokinetic).

#### 7.2.1.2. Derived Pharmacokinetic Parameters

The itraconazole and hydroxy-itraconazole plasma pharmacokinetic parameters listed below will be calculated in the same manner as nemiralisib pharmacokinetic parameters – see Section 7.1.1.2.

| Parameter | Parameter Description |
|---|---|
| AUC(0-∞) | Area under the concentration-time curve from zero time (pre-dose) extrapolated to infinite |
| | time. $AUC(0-\infty) = AUC(0-t) + C(t)/\lambda z$ . |
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration |
| %AUCex | Percentage of AUC(0-∞) obtained by extrapolation |
| Cmax | Maximum observed plasma concentration |
| tmax | Time to Cmax |
| t <sub>½</sub> | Apparent terminal half-life. $t_{1/2} = ln2/\lambda z$ |

#### NOTES:

- Additional parameters may be included as required.
- λz is the terminal phase rate constant

## 7.2.2. Summary Measure

The parameters for treatment comparisons are AUC(0- $\infty$ ), AUC(0-t), Cmax, tmax and  $t_{\frac{1}{2}}$  for both itraconazole and hydroxy-itraconazole.

#### 7.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

## 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed. Subjects with greater than 20% extrapolated AUC( $0-\infty$ ) will be flagged.

No formal statistical analysis will be performed.

## 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 8: List of Data Displays.

## 8.2. Adverse Events of Special Interest Analyses

Post-inhalation cough immediately following dosing is an adverse event of special interest (AESI). This will be captured if a participant reports it as an AE. The details of the planned displays are provided in Appendix 8: List of Data Displays.

## 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 8: List of Data Displays.

## 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 8: List of Data Displays.

# 9. PHARMACOKINETIC (POPPK)/ PHYSIOLOGICALLY-BASED PK (PBPK) ANALYSES

The study has been designed to capture the NCA pharmacokinetics of nemiralisib alone and when in the presence of itraconazole, to measure the effect, if any, on nemiralisib exposure. If the effect on nemiralisib exposure is large (increased AUC exposure due to markedly decreased clearance) then the sampling regimen may not be adequate for estimation of AUC( $0-\infty$ ) and a population PK or PBPK approach will be used to estimate AUC( $0-\infty$ ) of nemiralisib when in the presence of itraconazole. In such case, a separate CPMS RAP will be generated to describe the modelling work prospectively.

## 9.1. Statistical Analyses / Methods

A summary of the planned potential population pharmacokinetic analyses are outlined below:

- Drug nemiralisib concentration-time data will be subjected to nonlinear mixed effects modelling using the program NONMEM to develop a population PK model or a PBPK approach where more appropriate.
- o Individual post-hoc estimated PK parameters will be summarised descriptively.
- To support this analysis a PopPK dataset will be generated.

## 10. REFERENCES

GlaxoSmithKline Document Number 2017N347248\_00 Study ID 206874. A single centre, open label, one sequence, cross-over study to evaluate the effect of itraconazole on the pharmacokinetics of single inhaled doses of nemiralisib in healthy subjects. Report Date 12-DEC-2017.

## 11. APPENDICES

## 11.1. Appendix 1: Schedule of Activities

## 11.1.1. Protocol Defined Schedule of Events

Table 1 Screening and Follow-up

| Procedure | Screening (up to 21 days before Day 1) | Follow-up (within 5-10 days of last dose itraconazole) | Notes |
|---|---|---|---|
| Informed consent | X | | |
| Demography | X | | |
| Inclusion and exclusion criteria | Х | | |
| Past and current medical conditions | Х | | |
| Medical history (includes substance usage) | Х | | Substances: Drugs, Alcohol, tobacco and caffeine |
| Physical examination | Х | Х | Full examination (including height and weight) at screening, brief examination at follow-up |
| Vital signs | Х | | Triplicate |
| 12-lead ECG | Х | X | Triplicate |
| FEV <sub>1</sub> and FVC | X | | Triplicate |
| Laboratory assessments (hematology and clinical chemistry) | Х | Х | |
| Urinalysis | Х | | |
| HIV, Hepatitis B and C screening | Х | | If test otherwise performed within 3 months prior to first dose of study treatment, testing at screening is not required |
| Alcohol breath test & drug screen | Х | | Includes urine cotinine test |

2018N365720\_00 206874

| Procedure | Screening (up to 21 days<br>before Day 1) | Follow-up (within 5-10 days of last dose itraconazole) | Notes |
|---|---|---|---|
| SAE review | X | X | |
| AE review | | X | |

ECG: Electrocardigram, FEV1: Forced expiratory volume in 1 second, FVC: Forced vital capacity, HIV: Human immunodeficiency virus, AE: Adverse event, SAE: Serious adverse event.

Table 2 Period 1

| | | | Treatm | ent Peri | od Days | | | Notes |
|---|---|---|---|---|---|---|---|---|
| Procedure | -1 | 1 | 2 | 3 | 4 | 5 | 6 | |
| Admission | Χ | | | | | | | |
| Discharge | | | | | | | Χ | |
| Alcohol breath test & drug screen | Χ | | | | | | | Includes urine cotinine test |
| Laboratory assessments (hematology, clinical chemistry and urinalysis) | Х | | | | | | Х | Day −1 results to be reviewed before dosing on Day 1 |
| Brief physical examination | Х | | | | | | Х | |
| Inhaler (Ellipta™) training | Х | | | | | | | Training conducted by reviewing the Patient Information Leaflet with the participant. Additional training may be conducted at the discretion of the investigator. |
| FEV <sub>1</sub> | Χ | | | | | | | Triplicate. |
| 12-lead ECG | | Х | | | | | Х | Single measurement. Pre-dose on Day 1. |
| Vital signs | | Х | | | | | Х | Single measurement. Pre-dose on Day 1. |
| Study treatment (nemiralisib) | | Х | | | | | | |
| Pharmacokinetic (PK) (nemiralisib) | | Х | Х | Х | Х | Х | Χ | pre-dose, and 5 min, 30 min, 2 h, 6 h, 12 h, 24 h, 48 h, 72 h, 96 h and 120 h post-dose |
| AE review | | ←========→ | | ==> | | | | |
| SAE review | Х | <del>(====================================</del> | | | | | ==> | |
| Concomitant medication review | Χ | <del>(==</del> | | ===== | | | ==> | |

Table 3 Period 2

| | | | | | Trea | tment l | Period | Notes | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | |
| Admission | Χ | | | | | | | | | | | | |
| Discharge | | | | | | | | | | | | Х | |
| Alcohol breath test & drug screen | Х | | | | | | | | | | | | Includes urine cotinine test |
| Brief physical examination | Χ | | | | | | | | | | | Х | |
| Laboratory assessments (hematology, clinical chemistry and urinalysis) | Х | | | | | | | | | | Х | | Pre-dose at all timepoints. Day -1 results to be reviewed before dosing on Day 1. |
| Clinical chemistry only | | | Х | | Х | | Х | | Х | | | | Pre-dose at all timepoints. Day 4 results to be reviewed before itraconazole dosing on Day 5. |
| 12-lead ECG | | Х | х | | Х | | Х | | Х | | х | | Single measurement. Pre-dose and 3h post-dose (itraconazole) on Day 1. Pre-dose at all other timepoints, Day 4 results to be reviewed before itraconazole dosing on Day 5. |
| Vital signs | | Х | Χ | | Х | | Х | | Х | | Х | | Single measurement. Pre-dose at all timepoints |
| Study treatment (itraconazole) | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | Approx. 1 h post standard meal. |
| FEV <sub>1</sub> | | | | | Х | | | | | | | | Triplicate |
| Inhaler (Ellipta) training | | | | | Х | | | | | | | | Training conducted by reviewing the Patient Information Leaflet with the participant. Additional training may be conducted at the discretion of the investigator. |
| Study treatment (nemiralisib) | | | | | | Χ | | | | | | | 1 h post itraconazole administration. |
| PK (nemiralisib) | | | | | | Х | Х | Х | Х | Х | Х | Х | pre-dose, and 5 min, 30 min, 2 h, 6 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h and 144 h post-dose (nemiralisib) |

| | | | | | Trea | tment | Period | Notes | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | |
| PK (itraconazole + hydroxy-itraconazole) | _ | Х | | | | Х | х | L | _ | | | | Pre-dose, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h post-dose (itraconazole) on Day 1 Pre-dose, 30 min, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 24 h hours post-dose (itraconazole) on Day 5 |
| AE review | | + | ←======→ | | | | | | | | | | |
| SAE review | Х | + | ←======→ | | | | | | | | | | |
| Concomitant medication review | Х | + | | | | | ===== | | ===== | ===== | | $\rightarrow$ | |

- The timing and number of planned study assessments, including safety and pharmacokinetic assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments must be documented and approved by the relevant study team member and then archived in the sponsor and site study files, but will not constitute a protocol amendment. The Institutional review board (IRB)/ Independent ethics committee (IEC) will be informed of any safety issues that require alteration of the safety monitoring scheme or amendment of the Informed consent form (ICF).

# 11.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

## 11.2.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

• Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 11.2.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after study treatment start date (for that period) &amp; on or before nemiralisib treatment stop date (for that period) plus 10 days (5 times half life of nemiralisib).</li> <li>Study Treatment Start Date (for that period) ≤ AE Start Date ≤ Nemiralisib Treatment Stop Date (for that period) + 10 days.</li> <li>Where 'study treatment' start date (for that period) refers to the date of the first dose given in that period (i.e. nemiralisib for period 1 and itraconazole for period 2)</li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 11.3. Appendix 3: Data Display Standards & Handling Conventions

## 11.3.1. Reporting Process

| Software | |
|---|---|
| The currently sup | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Compound : GSK2269557/mid206874 | |
| Analysis Datasets | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version v3.2 &amp; ADaM IG<br/>Version 1.0.</li> </ul> | |
| Generation of RTF Files | |
| RTF files will be generated for the final reporting effort. | |

## 11.3.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in summary figures, summaries, statistical analyses and calculation of any derived parameters.
  - Actual relative time will be used in subject plots and for the derivation of PK parameters.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures.
- All unscheduled visits will be included in listings.

| Listings | |
|---|---|
| Since this is a single sequence study, there is no need to include 'Sequence' or 'Arm' in any of the listings. | |
| Descriptive Summar | Descriptive Summary Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

# 11.3.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | Pharmacokinetic Concentration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to PK IDSL Standards. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics and summarized graphical displays only. The number of values imputed will be included as a column in the summary tables. |
| NONMEM/Pop PK<br>File | Not applicable. |
| NONMEM/PK/PD<br>File | Not applicable. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameters to be<br>Derived by<br>Programmer | None |
| Pharmacokinetic Para | ameter Data |
| Is the 'NQ impacted PK Parameters' Rule Being Followed? | Yes, refer to Standards for Handling NQ Impacted PK Parameters. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

## 11.4. Appendix 4: Derived and Transformed Data

#### 11.4.1. General

#### **Multiple Measurements at One Analysis Time Point**

- The mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date within the period in question (in period 1 this will be the date of dosing with nemiralisib; in period 2 this will be the date of first dosing with itraconazole):
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 11.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard algorithms will be used for calculating age where birth date is imputed as:
  - Any subject with a missing day will have this imputed as day '15'.
  - Any subject with a missing date and month will have this imputed as '30th June'.
  - Birth date will be presented in listings as 'YYYY'.

#### Body Mass Index (BMI)

• Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Extent of Exposure**

- Number of days of exposure to each study drug will be calculated for each period based on the formula:
   Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were assigned treatment but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

#### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

• If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

## 11.4.3. Safety

#### **Adverse Events**

## AE Time Since First Dose (Days)

• If AE start date/time < date/time of first dose then

Time since first dose = date of first dose - AE start date

• If AE start date/time ≥ date/time of first dose then

Time since first dose = AE start date - date of first dose+1

- Missing if AE start date or date of first dose is missing.
- Note: First dose will be the date of dosing with nemiralisib in period 1 and the date of first dosing with itraconazole in period 2.

## AE Duration (Days)

- AE end date AE start date + 1
- Missing if AE start date or end date is missing.

## AE's of Special Interest

 Post-inhalation cough is an AE of special interest. The lower level term (LLT) to be included is "coughing after drug inhalation"

## 11.5. Appendix 5: Reporting Standards for Missing Data

## 11.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the last visit. |
| | <ul> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 11.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the output.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> <li>Data below the limit of quantification (BLQ) is not missing data and must be displayed as 'NQ (&lt; x)' where x is the lower limit of quantification, and included in all listings and summaries.</li> <li>Analysis will be performed on all available data and no imputation will be performed for missing data.</li> </ul> </li> </ul> |
| Outliers | <ul> <li>Any participants excluded from the summaries and/or statistical analyses because their<br/>values are considered outliers will be documented along with the reason for exclusion<br/>in the clinical study report.</li> </ul> |

## 11.5.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 2: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> <li>Note: start date and stop dates are defined as the first/last dose given in the period, regardless of whether it is nemiralisib or itraconazole.</li> </ul> </li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. |

| Element | Reporting Detail |
|---|---|
| | Consequently, time to onset and duration of such events will be missing. |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.6. Appendix 6: Values of Potential Clinical Importance

## 11.6.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | 35 | 60 |
| Hematocrit | % | Female | 35 | 60 |
| | | $\Delta$ from BL | <b>↓</b> 7.5 | |
| | g/L | Male | 130 | 180 |
| Haemoglobin | | Female | 120 | 170 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | 4.0 |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | 12.0 |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 600 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Total Protein | g/L | | 55 | 90 |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | µmol/L | | | 1.3 x ULN |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.7 | 1.25 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 155 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 11.6.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-----------------------------|-----------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTcF Interval | msec | ≤ 300 | ≥ 450 |
| Absolute PR Interval | msec | < 100 | >240 |
| Absolute Ventricular Rate | beats/min | <35 | >100 |
| Change from Baseline | | | |
| Increase from Baseline QTcF | msec | | >60 |

## 11.6.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------------|------------------------|--------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≤ 90 | ≥ 150 |
| Diastolic Blood Pressure | mmHg | ≤ 40 | ≥ 100 |
| Heart Rate | bpm | ≤ 35 | ≥ 100 |
| Respiration rate | breaths/min | ≤ 8 | ≥ 20 |
| Oral Temperature | °C | ≤ 35.5 | ≥ 37.5 |

# 11.7. Appendix 7: Abbreviations & Trade Marks

## 11.7.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| BLQ | Below Limit of Quantification |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PBPK | Physiologically Based PK |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |

| Abbreviation | Description |
|--------------|--------------------------------------------|
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| WNL | Windows Non-Linear |

## 11.7.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | |
|---------------------------------------------------------|---|
| None | 1 |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| NONMEM |
| SAS |
| WinNonlin |

## 11.8. Appendix 8: List of Data Displays

## 11.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.9 | |
| Pharmacokinetic | 2.1 to 2.10 | 2.1 to 2.10 |
| Safety | 3.1 to 3.10 | |
| Section | Listings | |
| ICH Listings | 1 to 32 | |
| Other Listings | 33 to 39 | |

## 11.8.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 9: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

## 11.8.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |
## 11.8.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1A | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.3. | Safety | ES4 | Summary of Participant Disposition at Each Study Period | ICH E3 | SAC |
| 1.4. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| Protoc | ol Deviation | I | | | - |
| 1.5. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popula | tion Analysed | | | | · |
| 1.6. | Enrolled | SP1A | Summary of Study Populations | IDSL<br>Total column only | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.7. | Safety | DM3 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.8. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC |
| 1.9. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |

### 11.8.5. Pharmacokinetic Tables

| Pharma | cokinetic: Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 2.1. | PK | PK01 | Summary of Nemiralisib Plasma Concentration-Time Data | Include footnote: 'Times are relative to dosing with nemiralisib'. | SAC |
| 2.2. | PK | PK01 | Summary of Itraconazole Plasma Concentration-Time Data (Period 2) | Still include treatment group as a variable Include footnote: 'Times are relative to dosing with itraconazole'. | SAC |
| 2.3. | PK | PK01 | Summary of Hydroxy Itraconazole Plasma Concentration-Time Data (Period 2) | Still include treatment group as a variable Include footnote: 'Times are relative to dosing with itraconazole'. | SAC |
| PK Para | ameter | | | | |
| 2.4. | PK | PK03 | Summary of Untransformed Derived Nemiralisib Plasma<br>Pharmacokinetic Parameters | Don't include 95% CI Include variable 'day' If any NC values, include n* column and add footnote: 'NOTE: n*=number of NC values'. Include footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.5. | PK | PK05 | Summary of Log-transformed Derived Nemiralisib Plasma<br>Pharmacokinetic Parameters | Include all parameters except %AUCex and tmax Include variable 'day'. If any NC values, include n* column and add footnote: 'NOTE: n*=number of NC values'. Include footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 2.6. | PK | PK03 | Summary of Untransformed Derived Itraconazole Plasma Pharmacokinetic Parameters (Period 2) | Don't include 95% CI. Still include treatment group as a variable. Include variable 'day'. If any NC values, include n* column and add footnote: 'NOTE: n*=number of NC values'. Include footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |
| 2.7. | PK | PK05 | Summary of Log-transformed Derived Itraconazole Plasma Pharmacokinetic Parameters (Period 2) | Include all parameters except %AUCex and tmax Still include treatment group as a variable. Include variable 'day' If any NC values, include n* column and add footnote: 'NOTE: n*=number of NC values'. Include footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.8. | PK | PK03 | Summary of Untransformed Derived Hydroxy Itraconazole Plasma Pharmacokinetic Parameters (Period 2) | Don't include 95% CI. Still include treatment group as a variable. Include variable 'day'. If any NC values, include n* column and add footnote: 'NOTE: n*=number of NC values'. Include footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |
| 2.9. | PK | PK05 | Summary of Log-transformed Derived Hydroxy Itraconazole Plasma Pharmacokinetic Parameters (Period 2) | Include all parameters except %AUCex and tmax Still include treatment group as a variable. Include variable 'day'. If any NC values, include n* column and add footnote: 'NOTE: n*=number of NC values'. Include footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |
| 2.10. | PK | Non Standard<br>PK_T1 | Summary of Statistical Analysis of Derived Nemiralisib Plasma AUC(0-inf) and Cmax | AUC(0-inf) and Cmax only (unless AUC(0-t) also analysed) Include MSE Include n* and footnote (in shell) if there are any NC values | SAC |

# 11.8.6. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 2.1. | PK | PK16b | Individual Nemiralisib Plasma Concentration-Time Plots (Linear and Semi-Log) by Subject | Separate plots per subject Add a horizontal dashed line at y-axis = 5 pg/mL and footnote: LLQ = 5 pg/mL | SAC |
| 2.2. | PK | PK24 | Individual Nemiralisib Plasma Concentration-Time Plots (Linear and Semi-Log) by Treatment Group | All subjects in the same treatment group on the same graph ("spaghetti plot"). Separate page per treatment. Add a horizontal dashed line at y-axis = 5 pg/mL and footnote: LLQ = 5 pg/mL | SAC |
| 2.3. | PK | PK17 | Mean Nemiralisib Plasma Concentration-Time Plots (Linear and Semi-Log) by Treatment Group | Add a horizontal dashed line at y-axis = 5 pg/mL and footnote: LLQ = 5 pg/mL | SAC |
| 2.4. | PK | PK18 | Median Nemiralisib Plasma Concentration-Time Plots (Linear and Semi-Log) by Treatment Group | Add a horizontal dashed line at y-axis = 5 pg/mL and footnote: LLQ = 5 pg/mL | SAC |
| 2.5. | PK | PK24 | Individual Itraconazole Plasma Concentration-Time Plots (Linear and Semi-Log) by Treatment Group (Period 2) | All subjects on the same graph ("spaghetti plot"). Still include treatment group Add a horizontal dashed line at y-axis = 2 ng/mL and footnote: LLQ = 2 ng/mL Add footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.6. | PK | PK19 | Mean (±SD) Itraconazole and Hydroxy-Itraconazole Plasma<br>Concentration-Time Plots (Linear and Semi-Log) by Treatment<br>Group (Period 2) | Both itraconazole and hydroxy- itraconazole on the same plot. +SD for itraconazole and -SD for hydroxy-itraconazole. Add a horizontal dashed line at y-axis = 2 ng/mL and footnote: LLQ = 2 ng/mL. Still include treatment group Add footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |
| 2.7. | PK | PK18 | Median Itraconazole and Hydroxy-Itraconazole Plasma<br>Concentration-Time Plots (Linear and Semi-Log) by Treatment<br>Group (Period 2) | Both itraconazole and hydroxy-<br>itraconazole on the same plot<br>Add a horizontal dashed line at y-axis =<br>2 ng/mL and footnote: LLQ = 2 ng/mL<br>Still include treatment group<br>Add footnote: 'Nemiralisib was<br>administered on Day 5 of Period 2.' | SAC |
| 2.8. | PK | PK24 | Individual Hydroxy-Itraconazole Plasma Concentration-Time Plots (Linear and Semi-Log) by Treatment Group (Period 2) | All subjects on the same graph ("spaghetti plot"). Still include treatment group Add a horizontal dashed line at y-axis = 2 ng/mL and footnote: LLQ = 2 ng/mL Add footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| PK Para | ameter | | | | |
| 2.9. | PK | PK28 | Individual Subject (+Geometric Mean and 90% CI) Derived Nemiralisib Plasma PK Parameters by Treatment Group | AUC(0-inf) and Cmax only (unless AUC(0-t) also analysed) Each parameter on a separate page All subjects to be indicated with an 'x' The two treatment groups on the x-axis Parameter values on a log scale on y-axis | SAC |
| 2.10. | PK | Non Standard<br>PK_F1 | Treatment Ratios (90% CIs) for Analysis of Derived Nemiralisib Plasma AUC(0-inf) and CMax | AUC(0-inf) and Cmax only (unless AUC(0-t) also analysed) All parameters on the x-axis of the same plot. Ratio on a log scale on y-axis | SAC |

### 11.8.7. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1CP / | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | Safety | AE1CP | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| Laborat | tory: Chemistry | 1 | | , | |
| 3.3. | Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 Include baseline values. Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2'. | SAC |
| Laborat | tory: Hematolo | gy | | , | |
| 3.4. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 Include baseline values. Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2'. | SAC |
| Laborat | tory: Urinalysis | | | | |
| 3.5. | Safety | UR3b | Summary of Urine Dipstick Results | ICH E3 Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2'. | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.6. | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC |
| 3.7. | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC |
| ECG | | | | | |
| 3.8. | Safety | EG1 | Summary of ECG Findings | IDSL Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2 | SAC |
| 3.9. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL Include baseline values. Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2'. | SAC |
| Vital Si | gns | | | | |
| 3.10. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 Include baseline values. Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2'. | SAC |

# 11.8.8. ICH Listings

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal | ICH E3 Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2. | SAC |
| 3. | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2. | SAC |
| 4. | Enrolled | CP_RA1x | Listing of Planned and Actual Treatments | IDSL Only include the following variables: Site ID, Subject, Period, Planned Treatment, Actual Treatment | SAC |
| Protoco | ol Deviations | l | | | |
| 5. | Safety | DV2A | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 6. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Popula | tions Analysed | | | | |
| 7. | Enrolled | SP3a | Listing of Participants Excluded from Any Population | ICH E3 | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 8. | Safety | DM4 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 9. | Safety | DM10 | Listing of Race | ICH E3 | SAC |
| Conco | mitant Medicati | ons | | | |
| 10. | Safety | CP_CM4 | Listing of Concomitant Medications | IDSL | SAC |
| Exposi | ıre | l | | | |
| 11. | Safety | EX4 | Listing of Nemiralisib Exposure Data | ICH E3 Include Period, Start Period Day (under study day), Stop Period Day (under study day). Don't include Cumulative Dose. Dosing Frequency = 'OD' | SAC |
| 12. | Safety | EX4 | Listing of Itraconazole Exposure Data | ICH E3 Include Period, Start Period Day (under study day), Stop Period Day (under study day), Cumulative Dose Dosing Frequency = 'OD' | SAC |
| Advers | e Events | | | | |
| 13. | Safety | AE9CP | Listing of All Adverse Events | ICH E3 Drop 'Maximum Grade' variable Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 16. | Safety | AE9CPA | Listing of Serious Adverse Events | ICH E3 Drop 'Maximum Grade' variable Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 17. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 18. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 Drop 'Maximum Grade' variable Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| Advers | e Events of Sp | ecial Interest | | | |
| 19. | Safety | AE9CP | Listing of Adverse Events Categorised as Post Inhalation Cough | Drop 'Maximum Grade' variable Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| Hepato | biliary (Liver) | | | | |
| 20. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC |
| 21. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | |
| 22. | Safety | LB6 | Listing of All Chemistry Data for Participants with Any Value of Potential Clinical Importance | ICH E3 Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 23. | Safety | LB6 | Listing of All Hematology Data for Participants with Any Value of Potential Clinical Importance | ICH E3 Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 24. | Safety | LB6 | Listing of Chemistry Values of Potential Clinical Importance | Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 25. | Safety | LB6 | Listing of Hematology Values of Potential Clinical Importance | Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 26. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 Include Treatment/Period and sort as for a crossover study. Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| ECG | | | | | |
| 27. | Safety | EG4 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL Include actual relative time. Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 28. | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance | IDSL Include actual relative time. Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 29. | Safety | EG6 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 30. | Safety | EG6 | Listing of Abnormal ECG Findings | IDSL Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| Vital Sig | gns | | | | |
| 31. | Safety | VS5 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| 32. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance | IDSL Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |

## 11.8.9. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| FEV <sub>1</sub> | | | | | |
| 33. | Safety | PFT10 | Listing of FEV1 and FVC Data | Include Treatment, Period, Day In terms of FEV1 and FVC, only need Max FEV1, Max FVC, % Predicted FEV1, % Predicted FVC Add Footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | SAC |
| PK Con | centration | | | | |
| 34. | PK | PK08 | Listing of Nemiralisib Plasma Concentration-Time Data | Add footnote: 'Times are relative to dosing with nemiralisib'. | SAC |
| 35. | PK | PK08 | Listing of Itraconazole Plasma Concentration-Time Data (Period 2) | Still include treatment group as a variable. Add footnote: 'Times are relative to dosing with itraconazole'. | SAC |
| 36. | PK | PK08 | Listing of Hydroxy Itraconazole Plasma Concentration-Time Data (Period 2) | Still include treatment group as a variable. Add footnote: 'Times are relative to dosing with itraconazole'. | SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Par | ameter | | | | |
| 37. | PK | PK14 | Listing of Derived Nemiralisib Pharmacokinetic Parameters | Include the variable 'day'. Flag AUC(0-inf) for subjects with >20%AUCex with a *. Add footnote:'*: Greater than 20% of AUC(0-inf) obtained by extrapolation'. | SAC |
| | | | | Add footnote: 'Nemiralisib was administered on Day 1 of Period 1 and Day 5 of Period 2.' | |
| 38. | PK | PK14 | Listing of Derived Itraconazole Pharmacokinetic Parameters (Period 2) | Include the variable 'day'. Still include treatment group as a variable. Flag AUC(0-inf) for subjects with | SAC |
| | | | | >20%AUCex with a *. Add footnote:'*: Greater than 20% of AUC(0-inf) obtained by extrapolation'. Add footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | |
| 39. | PK | PK14 | Listing of Derived Hydroxy Itraconazole Pharmacokinetic Parameters (Period 2) | Include the variable 'day'. Still include treatment group as a variable. Flag AUC(0-inf) for subjects with >20%AUCex with a *. Add footnote:'*: Greater than 20% of AUC(0-inf) obtained by extrapolation'. Add footnote: 'Nemiralisib was administered on Day 5 of Period 2.' | SAC |

### 11.9. Appendix 9: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request